CLINICAL TRIAL: NCT06136052
Title: The Effect of Kinesiophobia on Fear of Falling, Quality of Life and Physical Activity in Children With Headache
Brief Title: Kinesiophobia in Children With Headaches
Status: Completed | Type: Observational
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Lecturer, Muğla Sıtkı Koçman University
Other Study IDs: Kinezyofobivebasagrısı
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Headache; Kinesiophobia; Children
Keywords: headache; kinesiophobia; children
MeSH Terms: conditions — Headache; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Forms — All participants filled out a case evaluation form including demographic information, information about headache complaints, and scores of the questionnaire results. Participants completed the Tampa Kinesiophobia Scale (TKS) for kinesiophobia assessment. The International Fall Efficacy Scale (IFES) used in our study is a questionnaire consisting of 16 questions that provide information about the level of fear of falling during daily life activities. In our study, the visual analog scale (VAS), one of the most commonly used, oldest, and best validated scales, was used to measure pain intensity. The short form of the International Physical Activity Questionnaire (IPAQ)- consisting of seven questions- was used in our study. The Quality of Life Scale for Children (QoLSC) is a general quality of life scale that is widely used in research and evaluates the physical and psychosocial experiences of children between the ages of 2 and 18.

SUMMARY:
Introduction: Kinesiophobia is a common symptom associated with high levels of disability and has also been observed in patients with headache. However, the relationship between kinesiophobia and clinical factors in this population is unknown.

Objective: We aimed to investigate the relationship between kinesiophobia and fear of falling, quality of life, and physical activity in children with headache.

Methods: We included 127 children aged 6-18 years with headache complaints in our study. The Tampa Kinesiophobia Scale (TKS) was used to assess kinesiophobia, the International Falls Efficacy Scale (IFSES) was used to assess fear of falling, the International Physical Activity Questionnaire (IPAQ)- short form was used to measure physical activity, and the Quality of Life Scale for Children (QOLS) was used to assess quality of life. A visual analog scale (VAS) was used to assess pain intensity.

DETAILED DESCRIPTION:
Data for this cross-sectional study were collected from a convenient sample of patients aged 6-18 years with headache complaints who presented to a tertiary care pediatric neurology outpatient clinic between April 2022 and April 2023. The sampling size was determined as 88 at the beginning of the study and 127 patients were reached in our study. The inclusion criteria were determined as patients aged 6-18 years with headache complaints who applied to the pediatric neurology outpatient clinic of a training and research hospital, and the absence of any orthopedic, neurological, etc. disease that would prevent physical activity. The exclusion criteria were determined as having communication problems that would not allow evaluation and having a history of additional chronic diseases that would prevent physical activity. All participants filled out a case evaluation form including demographic information, information about headache complaints, and scores of the questionnaire results. Participants completed the Tampa Kinesiophobia Scale (TKS) for kinesiophobia assessment. The TKS consists of 17 questions inquiring about the increase in pain with movement, fear of injury, and avoidance of movement due to pain. The International Fall Efficacy Scale (IFES) used in our study is a questionnaire consisting of 16 questions that provide information about the level of fear of falling during daily life activities. In our study, the visual analog scale (VAS), one of the most commonly used, oldest, and best validated scales, was used to measure pain intensity. The short form of the International Physical Activity Questionnaire (IPAQ)- consisting of seven questions- was used in our study. In the questionnaire, respondents report the duration and frequency of their activities in the previous week. Measuring the quality of life of the individual with psychological tests is important for determining the quality of life of patients before and after treatment, evaluating the effectiveness and side effects of medical interventions, guiding health policies, and conducting medical research. The Quality of Life Scale for Children (QoLSC) is a general quality of life scale that is widely used in research and evaluates the physical and psychosocial experiences of children between the ages of 2 and 18, independent of illness.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years with headache complaints who applied to the pediatric neurology outpatient clinic
* absence of any orthopedic, neurological, etc. disease that would prevent physical activity.

Exclusion Criteria:

* having communication problems
* having a history of additional chronic diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Data for this cross-sectional study were collected from a convenient sample of patients aged 6-18 years with headache complaints who presented to a tertiary care pediatric neurology outpatient clinic between April 2022 and April 2023.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | 1 day
  Tampa Kinesiophobia Scale consists of 17 questions inquiring about the increase in pain with movement, fear of injury, and avoidance of movement due to pain.. The minimum score is 17 and the maximum score is 68. A score above 37 points indicates kinesiophobia.

SECONDARY OUTCOMES:
The International Fall Efficacy Scale (FES-I) | 1 day
  a questionnaire consisting of 16 questions that provide information about the level of fear of falling during daily life activities. Each question is scored from 1-4 (1= never worried, 2= a little worried, 3= quite worried, 4= very worried). The total score ranges from a minimum of 16 (no concern) to a maximum of 64 (extremely concerned). If the score is 24 or above, there is a fear of falling.
Visual Analog Scale | 1 day
  visual analog scale (VAS), one of the most commonly used, oldest, and best validated scales, was used to measure pain intensity. According to pain intensity, the scale is usually defined as "no pain" (0 points) and "as bad as possible" or "worst pain imaginable" (10 points). As the score increases, the pain intensity increases.
the International Physical Activity Questionnaire (IPAQ) | 1 day
  In the questionnaire, respondents report the duration and frequency of their activities in the previous week. The seven-item questionnaire provides information on time spent on sitting, walking, intermediate activities including sitting, and high-level activities. A score is calculated by multiplying the number of minutes, the number of days, and the MET value. For high and moderate physical activity and walking, values of 8 METs, 4 METs, and 3.3 METs are used, respectively. . The physical activity levels are classified as (< 600 MET-min/week), which is the physically inactive level (level I); (600-3000 MET- min/week), which is the level in medium-level (level II) and (> 3000 MET-min/week), which is the high physical activity level. The sitting score (sedentary behavior level) is calculated separately.
The Quality of Life Scale for Children (QoLSC) | 1 day
  Measuring the quality of life of the individual with psychological tests is important for determining the quality of life of patients before and after treatment, evaluating the effectiveness and side effects of medical interventions, guiding health policies, and conducting medical research.It takes a value between 0-100 points. As the score increases, the perception of quality of life increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Baykan Copurgolu, PhD(c), Principal Investigator — Kayseri University
Locations (1):
- Kayseri University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided